CLINICAL TRIAL: NCT00064935
Title: Utility of the Endometrial Biopsy in the Evaluation of the Luteal Phase
Brief Title: Endometrial Biopsy in Infertile Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Diagnostic
Other Study IDs: U01HD038997 (NIH); U01HD038997 (NIH); NICHD-0803
Record Dates: First submitted 2003-07-15; First posted 2003-07-16 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-05

CONDITIONS: Infertility
Keywords: Endometrium; Luteal phase; Endometrial biopsy
MeSH Terms: conditions — Infertility

INTERVENTIONS:
Procedure: Endometrial biopsy

SUMMARY:
When a woman becomes pregnant, the fertilized egg attaches itself to the lining of the uterus (endometrium). The endometrium is constantly changing throughout a woman's menstrual cycle in response to the female hormones estrogen and progesterone. The endometrium must have certain characteristics (be at a specific phase in its cycle) in order for the fertilized egg to successfully attach. Infertility may be caused by an "out of phase" endometrium (i.e., the endometrium doesn't have the right characteristics when the fertilized egg reaches it). The purpose of this study is to evaluate whether the endometrial biopsy is useful in predicting the potential for becoming pregnant and bearing a child.

DETAILED DESCRIPTION:
This study will evaluate the utility of the endometrial biopsy as a tool for the routine evaluation of the luteal phase of women presenting for infertility evaluation. The study will establish whether the mid-luteal or late-luteal phase is the most appropriate time to perform an endometrial biopsy. The study will be conducted through the multi-center Reproductive Medicine Network.

Women with a history of infertility will be age matched to fertile women (controls). Women will be randomized either to the mid-luteal phase (7 to 8 days post-ovulation) endometrial biopsy group or to the late-luteal phase (12 to 13 days post-ovulation) endometrial biopsy group. Endometrial specimens will be evaluated histologically by a "blinded" pathologist.

ELIGIBILITY:
Inclusion Criteria for Fertile Patients (controls)

* No history of involuntary primary or secondary infertility
* Willingness to discontinue hormonal contraceptives for 1 month prior to and through the duration of the study
* At least 1 child delivered within 24 months prior to study entry
* Most recent pregnancy resulting in a live birth (no interim spontaneous abortions)
* Tubal ligation within 24 months of study entry is acceptable if all other criteria are met

Inclusion Criteria for Infertile Patients

* History of primary or secondary infertility for a period of at least 12 months
* No hormonal treatments in the month preceding study entry
* No history of tubal ligation

Ages: 25 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 880
Dates: Start 1999-04; Study Completion 2002-02

CONTACTS AND LOCATIONS:
Overall Officials: Evan Myers, MD, MPH, Principal Investigator — Duke University Medical Center and Duke Clinical Research Institute
Locations (8):
- United States (8):
  - University of Alabama, Birmingham, Alabama
  - University of Colorado, Denver, Colorado
  - Wayne State University, Detroit, Michigan
  - University of Medicine and Dentistry, NJ, Newark, New Jersey
  - Pennsylvania State University, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas